CLINICAL TRIAL: NCT07284693
Title: Clinical Study Evaluating the Efficacy of Phenolic Complex k110-42 Therapy on Cognitive Functions of Children With Down Syndrome
Brief Title: Phenolic Complex k110-42 Therapy on Cognitive Functions in Down Children
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Haidi Sameh Ahmed Elassal, Resident, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ms.25.04.3157
Record Dates: First submitted 2025-11-30; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Functions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenolic complex k110-42 (Active Comparator): 900mg/kg oral once sachet for 6 month
  Interventions: Drug: Phenolic complex k110-42
- Neumentix (Placebo Comparator): Sachet once for 6 month
  Interventions: Drug: Neumentix

INTERVENTIONS:
Drug: Phenolic complex k110-42 — 900 mg/kg once oral in form of sachet for 6 month
  Arms: Phenolic complex k110-42
Drug: Neumentix — 0 mg/kg once sachet oral for 6 month
  Arms: Neumentix

SUMMARY:
The goal of this study is to evaluate the efficacy of phenolic complex k110-42 on cognitive function of children with Down syndrome

DETAILED DESCRIPTION:
Children with Down syndrome (DS) often face a variety of cognitive and developmental challenges. These challenges may include delays in speech, motor skills, and social-emotional development. Among these, difficulties with attention and focus are particularly prominent, making it harder for children with DS to participate in academic and everyday activities.

One promising avenue for improving cognitive function is the use of natural compounds with neuroprotective and cognitive-enhancing properties. The phenolic complex K110-42 (Neumentix), derived from the extract of spearmint, has garnered attention for its potential benefits in cognitive performance.

Specifically, polyphenols contained within the aqueous extracts from the Lamiaceae family could mechanistically account for the reported benefits on cognitive performance. Polyphenols found in aqueous extracts of spearmint such as salvianolic and rosmarinic acids have been shown to have anti-oxidant, anti-inflammatory, anti-acetylcholinesterase, and neuroprotective biological activity both in vitro and in vivo .

Phenolic offers a number of benefits on cognitive functions and it is plausible that its anti-inflammatory, antioxidant, anti-fibrotic effects, enhance attention, improving vascular endothelial functions and enhancement of metabolic performances. Because of the multiple functions, phenolic has direct effects on attention deficit in DS.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with Down syndrome (Non disjunction Trisomy 21) based on genetic testing .
* Age between 4-8 years old .
* Down syndrome children presented with difficulties in attention or focus as reported by parents or based on prior clinical assessments.

Exclusion Criteria:

* Parents' refusal.
* Down syndrome children with other significant developmental or neurological disorders (e.g., autism spectrum disorder, epilepsy).
* Patients with any chronic illness as liver or renal dysfunction; inflammatory diseases; autoimmune disease; cancer, acute cardiovascular event, eating disorders (anorexia, bulimia) or gastrointestinal disorders.
* Presence of hypersensitivity to spearmint or any components of Neumentix (Neumentix may increase kidney or liver damage if used in large amounts).
* Use of stimulant ADHD medication or cognitive-enhancing supplements .
* IQ test less than 55%.
* Patients with hypothyroidism.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive functions | At baseline before any intervention, at 3 month ,at 6 month
  Cognitive assessment will be assessed using Conners' Kiddie Continuous Performance Test (K-CPT).
Cognitive assessment will be assessed using the Wechsler Intelligence Scale for Children-Fourth Edition. | At baseline before any intervention , at 3 month , at 6 month

IPD SHARING:
Plan to Share IPD: No